CLINICAL TRIAL: NCT04771884
Title: Population Pharmacokinetics of Commonly Used Antimicrobial Agents in Children of Bacterial Meningitis With Augmented Renal Clearance
Status: Recruiting | Type: Observational
Sponsor: Shandong University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Wei Zhao, Professor; Head of department of clinical pharmacy and pharmacology, Shandong University
Other Study IDs: 2021-ARC-002
Record Dates: First submitted 2021-02-20; First posted 2021-02-25 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Bacterial Meningitis; Augmented Renal Clearance
MeSH Terms: conditions — Meningitis, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment(meropenem vancomycin ceftazidime ceftriaxone ceftizoxime linezolid): The use of antimicrobial agents depends on the clinical practice.
  Interventions: Drug: meropenem vancomycin ceftazidime ceftriaxone ceftizoxime linezolid

INTERVENTIONS:
Drug: meropenem vancomycin ceftazidime ceftriaxone ceftizoxime linezolid — The use of antimicrobial agents depends on the clinical practice

SUMMARY:
The investigator's purpose is to study the population pharmacokinetics of commonly used antimicrobial agents in children of bacterial meningitis with augmented renal clearance and assess dosage individualization feasibility.

DETAILED DESCRIPTION:
The investigator's purpose is to study the population pharmacokinetics of meropenem, vancomycin, ceftazidime, ceftriaxone, ceftizoxime and linezolid in children of bacterial meningitis with augmented renal clearance and assess dosage individualization feasibility. In this study, the investigator will detect drug concentration in both plasma and cerebrospinal fluid to construct population pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Children have been diagnosed with bacterial meningitis with augmented renal clearance (eGFR ≥ 160 mL/(min*1.73m2));
* Age: 2 months-18 years;
* Meropenem, vancomycin, ceftazidime, ceftriaxone, ceftizoxime and/ or linezolid used as part of regular treatment;
* Meropenem, vancomycin, ceftazidime, ceftriaxone, ceftizoxime and linezolid was administered intravenously.

Exclusion Criteria:

* Patients who die within the treatment cycle;
* Severe congenital malformation;
* Receive other systemic experimental drug therapy;
* Other factors that the researchers consider unsuitable for inclusion.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (2 months-18 years) of bacterial meningitis with augmented renal clearance
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
The peak plasma and cerebrospinal fluid drug concentration of meropenem，vancomycin，ceftazidime，ceftriaxone，ceftizoxime，linezolid. | at (5-10) minutes after intravenous administration
  To detect the peak plasma and cerebrospinal fluid drug concentration of meropenem，vancomycin，ceftazidime，ceftriaxone，ceftizoxime，linezolid after intravenous administration.
The random plasma and cerebrospinal fluid drug concentration of meropenem，vancomycin，ceftazidime，ceftriaxone，ceftizoxime，linezolid. | at (0.5-10) hours after intravenous administration
  To detect the random plasma and cerebrospinal fluid drug concentration of meropenem，vancomycin，ceftazidime，ceftriaxone，ceftizoxime，linezolid after intravenous administration.
The trough plasma and cerebrospinal fluid drug concentration of meropenem，vancomycin，ceftazidime，ceftriaxone，ceftizoxime，linezolid. | at 1-2 hours before the next administration
  To detect the trough plasma and cerebrospinal fluid drug concentration of meropenem，vancomycin，ceftazidime，ceftriaxone，ceftizoxime，linezolid after intravenous administration.

SECONDARY OUTCOMES:
clinical response | Through study completion, an average of 14 days
  Blood routine examination, cerebrospinal fluid routine examination and infection indicators (C-reaction protein, procalcitonin)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China